CLINICAL TRIAL: NCT03788707
Title: Performance of CO2 Changes to Predict Fluid Responsiveness in Spontaneously Breathing Volunteers
Brief Title: Capnogram and Fluid Responsiveness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19. The study was never started.
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor. Department of Anesthesiology, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1368341
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy; Blood Pressure

STUDY DESIGN:
Intervention Model Description: Volunteers will lay flat with a face mask breathing room air while expired CO2 is measured. After 30 seconds, legs will be passively raised for 3 minutes. Changes in expired CO2 before and after leg raising will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive leg raising (Experimental): Passive leg raising for 3 minutes after 20 seconds of lying flat
  Interventions: Other: Passive leg raising

INTERVENTIONS:
Other: Passive leg raising — After 30 seconds of lying flat, volunteers will have passive leg raising to 45 degrees. Expired CO2 will be measured via a face mask before and after leg raising.

SUMMARY:
Predicting fluid responsiveness in critically ill patients is of paramount importance. It can help define an adequate fluid balance. Overzealous fluid administration is poorly tolerated and has been associated with poor outcomes but so has insufficient administration. Currently available predictors of fluid responsiveness rely on invasive monitors and require patients to be on mechanical ventilation. It is thus important to develop non invasive novel methods to assess fluid responsiveness to provide an accurate management for a favorable outcome. We propose a readily available non-invasive method that relies on improvement of the ventilation perfusion mismatch as recorded by end tidal CO2.

Ventilation of physiologic dead space is part of a spectrum of mismatch between ventilation and perfusion of the lungs. The extent of pulmonary dead space varies depending on factors affecting pulmonary perfusion (e.g. pulmonary capillary hydrostatic pressure) and alveolar pressure (e.g. positive pressure ventilation). Compromised pulmonary capillary perfusion can lead to ventilation-perfusion mismatch in a patient with clear conductive airway and adequate alveolar oxygen pressure. Alveolar dead space results in decreased CO2 exchange that translates into lower levels of expired CO2.

Stroke volume of the right ventricle is a major determinant of the pulmonary capillary perfusion. Right ventricular cardiac output can be increased by passive lower limb elevation maneuver, which ultimately results in improvement of the ventilation to perfusion ratio. This effect leads to a higher participation of perfused (and ventilated) alveolar units in gas exchange and narrowing of the gradient between arterial and expired CO2 concentration. Performing a passive leg raising (PLR) maneuver leads to stroke volume enhancement in both healthy patients and in those experiencing hemodynamic instability. Responsiveness to PLR can be assessed by different methods including echocardiography and pulse pressure variation. Left ventricular cardiac output (LVCO) can be easily measured by transthoracic echo and be used as a surrogate of right ventricular preload changes. LVCO can thus be used to assess the fluid responsiveness of PLR and the effects of on end tidal CO2 that ensue.

We propose this study to test the hypothesis that expired CO2 is a reliable predictor of fluid responsiveness after performance of the PLR maneuver, based on the assumption that increasing right ventricular output causes a reduction of the ventilation to perfusion ratio, leading to increased levels of expired CO2. T

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years

Exclusion Criteria:

* Cardiovascular and respiratory disease reported by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Expired CO2 | 10 minutes
  Area under the curve of a capnogram tracing will be measured in milimiters

SECONDARY OUTCOMES:
Mean arterial pressure | 10 minutes
  Mean arterial pressure in mmHg measured by non invasive oscillometer
Heart rate | 10 minutes
  beats per minute measured by non invasive plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided